CLINICAL TRIAL: NCT05513196
Title: Bilateral Erector Spinal Plan Block in Postoperative Analgesia After Total Abdominal Hysterectomy: An Observational Study
Brief Title: Bilateral Erector Spinal Plan Block in Postoperative Analgesia After Total Abdominal Hysterectomy
Status: Completed | Type: Observational
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Engin Çetin, principal investigator, Kocaeli University
Other Study IDs: 2021-ESP
Record Dates: First submitted 2021-11-23; First posted 2022-08-24 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-11

CONDITIONS: Postoperative Pain
Keywords: postoperative pain; total abdominal hysterectomy; erector spinae plan block; morphine; visuel analog scale
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ESPB Group: Erector spinae plane block performed group.
  Interventions: Procedure: Erector spinae plane block (ESPB)
- Control Group: Control group.

INTERVENTIONS:
Procedure: Erector spinae plane block (ESPB) — Bilateral erector spinae plane block will be performed with 20 mL, 0.25% bupivacaine at T9 level preoperatively.
  Groups: ESPB Group

SUMMARY:
The importance of effective postoperative pain management is well known. Overall, for total abdominal hysterectomy operations are related with severe postoperative pain. The undesired effects of pain can be prevented with multimodal analgesia for the patient. Many regional anesthesia techniques can be preferred for total abdominal hysterectomy. The aim of this study is to investigate postoperative analgesia effect of erector spina plane block for total abdominal hysterectomy.

DETAILED DESCRIPTION:
Postoperative pain, which starts with tissue damage as a result of surgical procedures, gradually decreases with wound healing and ends. Pain due to tissue damage is an acute pain that varies in severity according to its size and region. It creates physiopathological changes in many organs and tissues and has negative effects on systems. This situation causes serious postoperative morbidity and mortality in patients. For these reasons, postoperative pain control is very important. Inadequate pain control can cause acute pain to turn into chronic pain. The occurrence of pain in the diseased area before the operation, the severity of surgical tissue damage, environmental, psychological and genetic factors increase the rate of development of chronic pain.

Multimodal analgesia in postoperative pain management is a strategy that combines different analgesic methods to provide more effective analgesia and to reduce side effects. Compared to monotherapy, less dose requirement and better pain management are targeted thanks to the additive and synergistic effect of different analgesic drugs. Thanks to this reduced dose, the incidence of drug-related side effects in patients is also reduced.

Erector spina plan block (ESPB) is a new regional anesthesia method used especially in abdominal and thoracic surgeries. It was first described by Forero et al. for the treatment of thoracic neuropathic pain. ESP block in 2017 and 2018; Many case reports for analgesic purposes in cervical, thoracic, abdominal and pelvic pain have been published, but detailed clinical studies have not been found. Since then, it has been considered that this interfascial plane block can be applied as an alternative to the neuraxial block for certain surgeries.

Under the guidance of ultrasonography, regional anesthesia applications can be performed more safely, easily and effectively than methods such as electrical stimulation and loss of resistance based on the determination of superficial landmarks. Uncertainty about the relationship of the needle with the surrounding tissue in peripheral nerve blocks performed with the traditional blind method causes a higher risk of failure and complication of the application. For this reason, Erector spina plan blocks made in our clinic are performed under ultrasound guidance. Complication due to erector spina plane block (pneumothorax) was reported in only two articles. There is also a report in the literature reporting that lower thoracic erector spina plane block causes involuntary motor block. However, it is stated that the possible complications associated with the block may be due to the failure of the technique.

The erector spina plane block technique consists of an injection of 20 mL of 0.25% bupivacaine, guided by USG, between the erector spinae muscle and the transverse process below it. The procedure is performed after the patient is seated, in the prone position, or in the lateral decubitus position and the target vertebral level has been defined. A high frequency linear USG probe is placed 3 cm lateral to the spinous process. On the hyperechoic transverse process, hypoechoic M.latissimus dorsi and M.rector spina are defined. The needle is then advanced from cephal to caudal or from caudal to cephalad until it remains in the interfascial plane. The correct position of the needle is confirmed by observing intramuscular diffusion of the drug following bupivacaine injection.

In the studies, the effectiveness of the erector spina plan block was controlled with the Visual Pain Scale (VAS) in the postoperative period. Therefore, in our study, we evaluated the effectiveness of postoperative pain with VAS. In our study, the patients in the control group will be those who did not undergo the block procedure. There is a 10 cm long line drawn horizontally on the Visual Pain Scale. The left end of this line represents no pain (VAS 0), and the other end represents the most severe pain imaginable (VAS 10). The patient is asked to mark a point on this 10 cm line according to the severity of the pain at that moment.

In our clinic, the efficacy of erector spina plane block has been demonstrated in studies performed in various surgeries. These studies include cholecystectomy, thoracic surgery, breast surgery, etc. made in operations. It has been shown in the literature that erector spina plane block is also effective in total abdominal hysterectomy operation. In this study, we aimed to show the effectiveness of the erector spina plane block, which is routinely applied in our clinic to prevent postoperative pain after total abdominal hysterectomy operations.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-2 patients
* patients undergo elective total abdominal hysterectomy

Exclusion Criteria:

* patient refusal
* ASA 3-4
* obesity (body mass index >35 kg/m2)
* infection of the skin at the site of needle puncture area patients
* with known allergies to any of the study drugs
* coagulopathy

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who undergo elective total abdominal hysterectomy surgery
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | Postoperative 24th hour
  Morphine consumption (mg) of patients with patient controlled analgesia device
Visuel analog scale | Postoperative 24th hour
  visuel analog scale of patients

CONTACTS AND LOCATIONS:
Overall Officials: engin MD çetin, Principal Investigator — Kocaeli Universty
Locations (1):
- Kocaeli University, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ivanusic J, Konishi Y, Barrington MJ. A Cadaveric Study Investigating the Mechanism of Action of Erector Spinae Blockade. Reg Anesth Pain Med. 2018 Aug;43(6):567-571. doi: 10.1097/AAP.0000000000000789. PMID 29746445
- [Background] Hamed MA, Goda AS, Basiony MM, Fargaly OS, Abdelhady MA. Erector spinae plane block for postoperative analgesia in patients undergoing total abdominal hysterectomy: a randomized controlled study original study. J Pain Res. 2019 Apr 30;12:1393-1398. doi: 10.2147/JPR.S196501. eCollection 2019. PMID 31118757
- [Result] De Cassai A, Geraldini F, Carere A, Sergi M, Munari M. Complications Rate Estimation After Thoracic Erector Spinae Plane Block. J Cardiothorac Vasc Anesth. 2021 Oct;35(10):3142-3143. doi: 10.1053/j.jvca.2021.02.043. Epub 2021 Feb 20. No abstract available. PMID 33731296
- See also: erector spinae plane block images — http://www.nysora.com/erector-spinae-plane-block